CLINICAL TRIAL: NCT05047848
Title: Clinical Study of Chidamide Combined With Fulvestrant in the Treatment of Hormone Receptor-positive Advanced Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Tao Sun, Director, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C18
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide + fulvestrant (Experimental)
  Interventions: Drug: Chidamide; Drug: Fulvestrant

INTERVENTIONS:
Drug: Chidamide — chidamide 30mg orally，Biw
Drug: Fulvestrant — Fulvestrant 500mg i.m. injections every 28 days (Cycle n Day 1) with 1 additional dose on Day 15 of Cycle 1

SUMMARY:
This is a Open-label study of chidamide in combination with fulvestrant for the treatment of postmenopausal women with hormone receptor positive, Her2 negative, advanced breast cancer who have received no or only one line of endocrine therapy for advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. women aged ≥ 18 years, histologically or cytologically confirmed HR positive (ER expression ≥ 10%, PR positive or negative), HER2 negative breast cancer patients;
2. before enrollment for unresectable locally advanced or metastatic breast cancer, and at least one measurable lesion or no measurable lesion and bone metastasis alone patients;
3. For locally advanced or metastatic breast cancer, no previous endocrine therapy or first-line endocrine therapy, and no previous use of CDK4/6 inhibitors. Specifically, it includes the following conditions:

   Cohort 1: (neo) recurrence > 12 months after the end of adjuvant endocrine therapy, and without any rescue therapy · newly diagnosed advanced breast cancer without any rescue therapy Cohort 2: (neo) recurrence during or ≤ 12 months after the completion of adjuvant endocrine therapy, and without any rescue therapy · recurrence > 12 months after the completion of adjuvant endocrine therapy, and progression by first-line endocrine therapy · newly diagnosed advanced breast cancer and progression by first-line endocrine rescue therapy
4. Cohort 1 without previous chemotherapy for advanced breast cancer; Cohort 2 with ≤ 1 previous chemotherapy for advanced breast cancer;
5. no brain metastasis or asymptomatic brain metastasis;
6. ECOG score 0-1;
7. Absolute neutrophil count ≥ 1.5 × 109/L, platelet ≥ 100 × 109/L, hemoglobin ≥ 90 g/L;
8. Expected survival time ≥ 3 months;
9. Voluntarily participate in this clinical trial, sign the written informed consent;

Exclusion Criteria:

1. no measurable lesions (except bone metastases alone), such as pleural or pericardial exudates, ascites, etc.
2. Patients who have undergone major surgical procedures or significant trauma before enrollment, or are expected to undergo major surgical treatment
3. Patients who have previously been treated with CDK4/6 inhibitors, fulvestrant or HDAC inhibitors (including romidepsin, vorinostat, berlistat, parabrestat), but have received 1 cycle (≤ 2 times, on d1, d15, respectively) of fulvestrant within 28 days (before enrollment) are allowed
4. Known history of allergy to the drug components of this protocol
5. Meningeal metastasis before enrollment
6. Uncontrollable serosal effusion
7. Active infection [an active bacterial, viral, fungal, mycobacterial, parasitic or other infection (excluding fungal infections of the nail bed) within 4 months prior to Screening or any major infectious event requiring intravenous antibiotics, or targeted antiviral therapy, or hospitalization], or persistent fever within 14 days prior to Screening
8. a history of immunodeficiency, including HIV test positive, or suffering from other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
9. according to the investigator's judgment, there are serious hazards to the patient's safety, or affect the patient to complete the study of concomitant diseases (such as: severe hypertension, diabetes, thyroid disease, active infection, etc.);
10. History of definite neurological or psychiatric disorders, including epilepsy or dementia
11. Subjects who, in the opinion of the investigator, are not suitable for the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-06-18 (Estimated); Study Completion 2023-09-18 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 26 months
  Overall response rate (ORR) is defined as the proportion of patients with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 26 months
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause.
Overall Survival (OS) | Up to approximately 58 months
  Time from date of randomization to the date of death from any cause.
Clinical Benefit Rate (CBR) | Up to approximately 26 months
  Clinical benefit rate (CBR), defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1.
Duration of Response (DOR) | Up to approximately 26 months
  Time from the first documented response (CR or PR) to the first documented progression or death due to underlying cancer as defined in RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Liangning Tumor Hospital &Institute, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided